CLINICAL TRIAL: NCT02679573
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Comparator-Controlled Study to Evaluate the Safety and Efficacy of Intravenous to Oral Delafloxacin in Adult Subjects With Community-Acquired Bacterial Pneumonia
Brief Title: Study to Compare Delafloxacin to Moxifloxacin for the Treatment of Adults With Community-acquired Bacterial Pneumonia
Acronym: DEFINE-CABP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Melinta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ML-3341-306; 2015-003026-14 (EudraCT Number)
Record Dates: First submitted 2016-01-27; First posted 2016-02-10 (Estimated); Results first posted 2020-02-27 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Community Acquired Bacterial Pneumonia
Keywords: Pneumonia
MeSH Terms: conditions — Pneumonia | interventions — delafloxacin; Moxifloxacin; Linezolid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Delafloxacin (Experimental): IV delafloxacin with potential to switch to oral delafloxacin
  Interventions: Drug: Delafloxacin
- Moxifloxacin/Linezolid (Active Comparator): IV moxifloxacin with potential to switch to oral moxifloxacin, and potential to switch moxifloxacin to IV linezolid for confirmed MRSA
  Interventions: Drug: Moxifloxacin; Drug: Linezolid

INTERVENTIONS:
Drug: Delafloxacin — Antibacterial agent, 300 mg IV, Q12H for at least 6 doses with potential to switch to 450 mg oral tablet, Q12H for up to 20 doses total
  Other Names: RX-3341
  Arms: Delafloxacin
Drug: Moxifloxacin — Antibacterial Agent, 400 mg IV, Q24H for at least 3 doses with potential to switch to 400 mg oral over-encapsulated tablet, Q24H for up to 10 doses total
  Other Names: Avelox
  Arms: Moxifloxacin/Linezolid
Drug: Linezolid — Antibacterial Agent, at local investigator discretion, subjects in the moxifloxacin arm with confirmed MRSA can switch to linezolid 600 mg IV Q12H for all remaining doses
  Other Names: Zyvox
  Arms: Moxifloxacin/Linezolid

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of delafloxacin compared to moxifloxacin in the treatment of adult patients with community-acquired pneumonia.

DETAILED DESCRIPTION:
The purpose of this study is to determine if delafloxacin, an investigational drug, is safe and effective in the treatment of community-acquired bacterial pneumonia compared with moxifloxacin, or linezolid in the case of confirmed MRSA.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18 years of age or older
2. Evidence of acute onset of CABP with 2 or more of the following symptoms (new or worsening)

   * Cough
   * Production of purulent sputum consistent with bacterial infection
   * Difficulty breathing
   * Chest pain due to pneumonia

   AND have at least 2 of the following findings:
   * Fever (oral temperature >38.0°C)
   * Hypothermia (oral temperature <35.0°C)
   * Tachycardia (heart rate >100 beats/min)
   * Tachypnea (respiratory rate >18 breaths/min)

   AND have at least 1 of the following findings:
   * Hypoxemia (oxygen saturation <90% or PaO2 < 60 mmHg) on room air or with subject's baseline (pre-CABP under study) supplemental oxygen
   * Clinical evidence of pulmonary consolidation and/or presence of pulmonary rales
   * An elevated white blood cell count (WBC) >10,000/mm3 or 15% immature neutrophils (bands), regardless of total peripheral WBC count or leukopenia with WBC <4500/mm^3
3. Presence of lobar, multilobar, or patchy parenchymal infiltrate(s) consistent with acute bacterial pneumonia on a pulmonary imaging study within 48 hours before the first dose of study drug
4. PORT risk class of II to V (PSI score >50)
5. Must be a suitable candidate for possible IV to oral switch antibiotic therapy and must also be able to swallow large tablets/capsules intact without crushing

Exclusion Criteria:

1. A medical history of significant hypersensitivity or allergic reaction to antibiotics of the quinolone or oxazolidinone class or study drug excipients according to the investigator
2. Any infection expected to require other systemic antibiotics in addition to study drug
3. Receipt of systemic antibiotic therapy in the 7 days before enrollment unless 1 of the following is documented:

   * Received at least 48 hours of antibiotic therapy for CABP and clinic notes document treatment failure (i.e., not by patient history or pulmonary imaging alone) with new or worsening symptoms while on pre-study therapy
   * Received 1 dose of a single, potentially effective, short-acting antibacterial drug or drug regimen for CABP within 24 hours before enrollment (limited to 25% of enrolled patients)
4. Respiratory infection confirmed or suspected to be secondary to hospital-acquired or ventilator-associated pneumonia OR requires treatment in an intensive care setting, OR requires mechanical ventilation
5. Current or suspected diagnosis of viral, fungal, or aspiration pneumonia, noninfectious causes of pulmonary infiltrates, lung cancer, cystic fibrosis, tuberculosis, empyema (not including sterile parapneumonic effusions)
6. Known anatomical or pathological bronchial obstruction OR history of bronchiectasis OR GOLD Stage 4 COPD OR history of post obstructive pneumonia
7. Severely compromised immune system
8. Known history of Child-Pugh Class B or C liver disease
9. History of post-antibiotic colitis within last 3 months
10. Other exclusions include those described in the safety label for drugs in the quinolone and/or oxazolidinone classes such as QT prolongation, proarrhythmic conditions, concomitant use of drugs known to cause QT prolongation, peripheral neuropathy, tendon disorders, history of myasthenia gravis, liver disease, severe renal disease, seizures and concomitant use of MAO A or B inhibitor agents and adrenergic serotonergic agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 860 (Actual)
Dates: Start 2016-12-14 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-08-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sue Cammarata, MD, Study Director — Melinta Therapeutics, Inc.
Locations (89):
- United States (24):
  - Melinta 306 Study Site, Montgomery, Alabama
  - Melinta 306 Study Site, Newark, Delaware
  - Melinta 306 Study Site, Coral Gables, Florida
  - Melinta 306 Study Site, DeBary, Florida
  - Melinta 306 Study Site, DeLand, Florida
  - Melinta 306 Study Site, Fort Myers, Florida
  - Melinta 306 Study Site, Miami, Florida
  - Melinta 306 Study Site, Louisville, Kentucky
  - Melinta 306 Study Site, Natchitoches, Louisiana
  - Melinta 306 Study Site, Baltimore, Maryland
  - Melinta 306 Study Site, Boston, Massachusetts
  - Melinta 306 Study Site, Burlington, Massachusetts
  - Melinta 306 Study Site, Saint Paul, Minnesota
  - Melinta 306 Study Site, St Louis, Missouri
  - Melinta 306 Study Site, Butte, Montana
  - Melinta 306 Study Site, Omaha, Nebraska
  - Melinta 306 Study Site, Newark, New Jersey
  - Melinta 306 Study Site, Buffalo, New York
  - Melinta 306 Study Site, Charlotte, North Carolina
  - Melinta 306 Study Site, Cleveland, Ohio
  - Melinta 306 Study Site, Dayton, Ohio
  - Melinta 306 Study Site, Rapid City, South Dakota
  - Melinta 306 Study Site, Franklin, Tennessee
  - Melinta 306 Study Site, Corsicana, Texas
- Argentina (3):
  - Melinta 306 Study Site, Buenos Aires
  - Melinta 306 Study Site, Córdoba
  - Melinta 306 Study Site, La Plata
- Bulgaria (4):
  - Melinta 306 Study Site, Pleven
  - Melinta 306 Study Site, Rousse
  - Melinta 306 Study Site, Sofia
  - Melinta 306 Study Site, Stara Zagora
- Colombia (5):
  - Melinta 306 Study Site, Barranquilla
  - Melinta 306 Study Site, Cali
  - Melinta 306 Study Site, Manizales
  - Melinta 306 Study Site, Medellín
  - Melinta 306 Study Site, Quindío
- Melinta 306 Study Site, Santo Domingo, Dominican Republic
- Melinta 306 Study Site, Tbilisi, Georgia
- Germany (2):
  - Melinta 306 Study Site, Leverkusen
  - Melinta 306 Study Site, Munich
- Hungary (6):
  - Melinta 306 Study Site, Budapest
  - Melinta 306 Study Site, Debrecen
  - Melinta 306 Study Site, Deszk
  - Melinta 306 Study Site, Miskolc
  - Melinta 306 Study Site, Nyíregyháza
  - Melinta 306 Study Site, Szombathely
- Latvia (3):
  - Melinta 306 Study Site, Daugavpils
  - Melinta 306 Study Site, Liepāja
  - Melinta 306 Study Site, Riga
- Melinta 306 Study Site, Lima, Peru
- Poland (4):
  - Melinta 306 Study Site, Chrzanów
  - Melinta 306 Study Site, Katowice
  - Melinta 306 Study Site, Lodz
  - Melinta 306 Study Site, Wroclaw
- Romania (4):
  - Melinta 306 Study Site, Brasov
  - Melinta 306 Study Site, Bucharest
  - Melinta 306 Study Site, Craiova
  - Melinta 306 Study Site, Timișoara
- Russia (5):
  - Melinta 306 Study Site, Arkhangelsk
  - Melinta 306 Study Site, Moscow
  - Melinta 306 Study Site, Saint Petersburg
  - Melinta 306 Study Site, Smolensk
  - Melinta 306 Study Site, Vsevolozhsk
- Serbia (4):
  - Melinta 306 Study Site, Belgrade
  - Melinta 306 Study Site, Kamenitz
  - Melinta 306 Study Site, Kragujevac
  - Melinta 306 Study Site, Niš
- Slovenia (2):
  - Melinta 306 Study Site, Golnik
  - Melinta 306 Study Site, Ljubljana
- South Africa (8):
  - Melinta 306 Study Site, Benoni
  - Melinta 306 Study Site, Chatsworth
  - Melinta 306 Study Site, Krugersdorp
  - Melinta 306 Study Site, Middelburg
  - Melinta 306 Study Site, Phoenix
  - Melinta 306 Study Site, Port Elizabeth
  - Melinta 306 Study Site, Pretoria
  - Melinta 306 Study Site, Worcester
- Spain (5):
  - Melinta 306 Study Site, Badalona
  - Melinta 306 Study Site, Barcelona
  - Melinta 306 Study Site, Madrid
  - Melinta 306 Study Site, Terrassa
  - Melinta 306 Study Site, Valencia
- Ukraine (7):
  - Melinta 306 Study Site, Dnipro
  - Melinta 306 Study Site, Kharkiv
  - Melinta 306 Study Site, Kyiv
  - Melinta 306 Study Site, Poltava
  - Melinta 306 Study Site, Vinnytsia
  - Melinta 306 Study Site, Zaporizhia
  - Melinta 306 Study Site, Zhytomyr

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 860 subjects were planned to be enrolled in the study but 859 are included in the ITT population. One subject mistakenly was randomized into the IXRS but did not provide informed consent; therefore, this subject was not included in the ITT population.
Groups:
- Delafloxacin: Delafloxacin: 300 mg IV, Q12H for at least 6 doses with potential to switch to 450 mg oral tablet, Q12H for up to 20 doses total
- Moxifloxacin/Linezolid: Moxifloxacin: 400 mg IV, Q24H for at least 3 doses with potential to switch to 400 mg oral over-encapsulated tablet, Q24H for up to 10 doses total
  Linezolid: At local investigator discretion, subjects in the moxifloxacin arm with confirmed MRSA can switch to linezolid 600 mg IV Q12H for all remaining doses
Period: Overall Study
Arm/Group | Delafloxacin | Moxifloxacin/Linezolid
Started | 431 | 428
Completed | 394 | 389
Not Completed | 37 | 39
Not completed — Adverse Event | 13 | 6
Not completed — Lack of Efficacy | 12 | 15
Not completed — Could not complete required study visits | 6 | 2
Not completed — Withdrawal by Subject | 2 | 9
Not completed — Death | 2 | 0
Not completed — Physician Decision | 2 | 4
Not completed — Lost to Follow-up | 0 | 3

BASELINE CHARACTERISTICS:
Population: ITT Population comprised all randomized subjects with a signed ICF. Subjects were analyzed according to the treatment arm to which they were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Delafloxacin | Moxifloxacin/Linezolid | Total
Number analyzed (Participants) | 431 | 428 | 859
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 228 | 249 | 477
  >=65 years | 203 | 179 | 382
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (16.06) | 59.3 (61.0) | 60.0 (16.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 180 | 175 | 355
  Male | 251 | 253 | 504
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 32 | 23 | 55
  Not Hispanic or Latino | 399 | 405 | 804
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 0 | 4
  Asian | 5 | 5 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 22 | 33 | 55
  White | 398 | 388 | 786
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  Colombia | 11 | 9 | 20
  Argentina | 12 | 8 | 20
  Romania | 30 | 29 | 59
  Hungary | 14 | 12 | 26
  United States | 1 | 5 | 6
  Ukraine | 84 | 84 | 168
  Russia | 38 | 42 | 80
  Spain | 10 | 14 | 24
  Latvia | 19 | 21 | 40
  Dominican Republic | 2 | 0 | 2
  Poland | 20 | 8 | 28
  South Africa | 30 | 41 | 71
  Georgia | 45 | 50 | 95
  Slovenia | 8 | 7 | 15
  Bulgaria | 33 | 25 | 58
  Serbia | 69 | 73 | 142
  Peru | 4 | 0 | 4
  Germany | 1 | 0 | 1
PORT Risk Class [Count of Participants; unit: Participants] — Pneumonia Patient Outcomes Research Team (PORT) Risk Class (I-V) determined using the Pneumonia Severity Index (PSI).
  PSI Score / PORT Risk Class / Risk:
  ≤70 / II / Low, 71-90 / III / Low, 91-130 / IV / Moderate, >130 / V / High. Retrieved from http://www.mdcalc.com/psi-port-score-pneumonia-severity-index-adult-cap/ (Fine MJ, Auble TE, Yealy DM, et al. A prediction rule to identify low-risk patients with community-acquired pneumonia. N Engl J Med. 1997;336:243-50.)
  Participants
    II | 54 | 57 | 111
    III | 258 | 260 | 518
    IV | 115 | 103 | 218
    V | 4 | 8 | 12

OUTCOME MEASURES:

1. Primary Outcome: Early Clinical Response
Description: Early clinical response defined as improvement in at least 2 of the following symptoms (as assessed by the investigator): chest pain, frequency or severity of cough, amount and quality of productive sputum, and difficulty breathing, and no worsening of the other symptoms in the ITT population. Symptom severity evaluated by the investigator on a 4-point scale: Absent (0), Mild (1), Moderate (2), Severe (3). Improvement defined as at least a 1-point decrease from baseline.
Time Frame: 96 (+/- 24) hours after the first dose of study drug
Population: ITT (intent-to-treat) Population is all the randomized patients with a signed Informed consent form. Subjects were analyzed according to the treatment arm to which they were randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Delafloxacin | Moxifloxacin/Linezolid
Number analyzed (Participants) | 431 | 428
Participants | 383 | 381
Statistical Analysis 1: Comparison: Delafloxacin vs Moxifloxacin/Linezolid; The null (H0) and alternative (Ha) hypotheses to be tested to establish the noninferiority of delafloxacin were: H0: Pd - Pm ≤ -0.125 Ha: Pd - Pm > -0.125 where Pd and Pm are the probabilities of the ECR for delafloxacin and moxifloxacin, respectively. The treatment difference (delafloxacin - moxifloxacin) were presented, and the Miettinen-Nurminen test, without stratification, was used for the 2 sided 95% CI on the difference in response rate; Test type: Non-Inferiority — Used on a normal approximation approach (Miettinen and Nurminen's Likelihood Score Test), 860 subjects in the ITT population provided a 90% power to assess non-inferiority of delafloxacin vs. moxifloxacin based on the following assumptions: (1) a rate of ECR for moxifloxacin therapy and delafloxacin of 77% and 74%, respectively; (2) 1 sided type I error (α) of 0.025; and (3) a non-inferiority margin of 12.5%; Difference in responder rates = -0.2, 95% CI 2-sided [-4.4 to 4.1] — Difference = Difference in responder rates (Delafloxacin treatment group minus Moxifloxacin treatment group). Confidence intervals are calculated using Miettinen and Nurminen method without stratification

2. Secondary Outcome: Early Clinical Response Plus Improvement in Vital Signs and no Worsening of the 4 Symptoms
Description: Early clinical response with the addition of improvement in vital signs and no worsening of the following 4 symptoms: chest pain, cough, productive sputum, and difficulty breathing in the ITT population. Symptom severity evaluated by the investigator on a 4-point scale: Absent (0), Mild (1), Moderate (2), Severe (3). Improvement defined as at least a 1-point decrease from baseline. Improvement in vital signs defined as a return to normal of any abnormal vital signs at baseline, and no worsening (ie, be abnormal) of any vital sign that was normal at baseline.
Time Frame: 96 (+/- 24) hours after the first dose of study drug
Population: ITT (intent-to-treat) Population is all randomized patients with a signed Informed consent form. Subjects were analyzed according to the treatment arm to which they were randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Delafloxacin | Moxifloxacin/Linezolid
Number analyzed (Participants) | 431 | 428
Participants | 227 | 184
Statistical Analysis 1: Comparison: Delafloxacin vs Moxifloxacin/Linezolid; The null (H0) and alternative (Ha) hypotheses to be tested to establish the noninferiority of delafloxacin were: H0: Pd - Pm ≤ -0.125 Ha: Pd - Pm > -0.125 where Pd and Pm are the probabilities of the ECR for delafloxacin and moxifloxacin, respectively. The treatment difference (delafloxacin - moxifloxacin) was presented, and the Miettinen-Nurminen test without stratification was used for the 2 sided 95% CI on the difference in response rate; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Difference in responder rates = 9.7, 95% CI 2-sided [3.0 to 16.3]

3. Secondary Outcome: Clinical Outcome at Test of Cure
Description: Clinical outcome (Success, Failure, or Indeterminate/missing) based on the investigator's assessment of the patient's signs and symptoms of infection in the ITT population.
Time Frame: 5 to 10 days after the last dose of study drug
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Delafloxacin | Moxifloxacin/Linezolid
Number analyzed (Participants) | 431 | 428
Participants
  Success | 390 | 384
  Failure | 21 | 21
  Indeterminate/Missing | 20 | 23
Statistical Analysis 1: Comparison: Delafloxacin vs Moxifloxacin/Linezolid; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Difference in responder rates = 0.8, 95% CI 2-sided [-3.3 to 4.8]

4. Secondary Outcome: Clinical Outcome at End of Treatment
Description: as for outcome 3
Time Frame: Up to 24 (+4) hours after the last dose of study drug
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Delafloxacin | Moxifloxacin/Linezolid
Number analyzed (Participants) | 431 | 428
Participants
  Success | 396 | 390
  Failure | 19 | 20
  Indeterminate/Missing | 16 | 18
Statistical Analysis 1: Comparison: Delafloxacin vs Moxifloxacin/Linezolid; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Difference in responder rates = 0.8, 95% CI 2-sided [-3.0 to 4.6]

5. Secondary Outcome: Microbiologic Response
Description: Microbiological response for subjects in the MITT set will be based on results of the baseline and follow-up cultures and susceptibility testing or serology.
Time Frame: 5 to 10 days after the last dose of study drug
Population: Microbiological ITT 1 (MITT-1) includes all subjects in the ITT population with a baseline bacterial pathogen identified that was known to cause CABP and against which the study drug had antibacterial activity.
Measure: Count of Participants; unit: Participants
Arm/Group | Delafloxacin | Moxifloxacin/Linezolid
Number analyzed (Participants) | 257 | 263
Participants | 231 | 235
Statistical Analysis 1: Comparison: Delafloxacin vs Moxifloxacin/Linezolid; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Difference in responder rates = 0.5, 95% CI 2-sided [-4.8 to 5.9]

6. Secondary Outcome: All-cause Mortality
Description: Time to all-cause Mortality was assessed on Day 28.
Time Frame: Day 28 (+/- 2 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Delafloxacin | Moxifloxacin/Linezolid
Number analyzed (Participants) | 431 | 428
Participants | 8 | 6
Statistical Analysis 1: Comparison: Delafloxacin vs Moxifloxacin/Linezolid; Test type: Other; p = 0.5951, Log Rank — The log-rank test was used to compare the time to all-cause mortality between the 2 treatment groups

ADVERSE EVENTS:
Time Frame: All adverse events reported or observed during the study will be recorded from the time that the subject is first administered double-blind study drug through the End of Treatment (5 - 10 days) or Test of Cure visit (5 - 10 days after last dose), whichever is later. All serious adverse events will be recorded from the time the subject or authorized representative signs the informed consent form through the Follow up visit (Day 28).
Description: Adverse Events are reported in the Safety Population which includes all randomized subjects who received at least 1 dose of study drug. Two subjects in the delafloxacin group and 1 subject in the moxifloxacin group were randomized, but did not receive any study drug.
Arm/Group | Delafloxacin | Moxifloxacin/Linezolid
All-Cause Mortality (participants affected / at risk) | 8/429 | 6/427
Serious Adverse Events (participants affected / at risk) | 23/429 | 20/427
Other Adverse Events (participants affected / at risk) | 40/429 | 30/427
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Delafloxacin (N=429) | Moxifloxacin/Linezolid (N=427)
Pneumonia (Infections and infestations) | 3 (3) | 1 (1)
Septic Shock (Infections and infestations) | 3 (4) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 1 (1)
Herpes zoster meningomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 0 (0)
Lung abscess (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Measles (Infections and infestations) | 0 (0) | 1 (1)
Oral Herpes (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal bacteremia (Infections and infestations) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 2 (2)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Sarcoidosis (Immune system disorders) | 1 (1) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Agranulocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Sudden death (General disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Vertebrobasilar insufficiency (Nervous system disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Delafloxacin (N=429) | Moxifloxacin/Linezolid (N=427)
Diarrhoea (Gastrointestinal disorders) | 20 (21) | 14 (14)
Transaminases increased (Investigations) | 13 (13) | 6 (6)
Headache (Nervous system disorders) | 8 (8) | 11 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2017-12-04): https://cdn.clinicaltrials.gov/large-docs/73/NCT02679573/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-02): https://cdn.clinicaltrials.gov/large-docs/73/NCT02679573/SAP_001.pdf